CLINICAL TRIAL: NCT05377918
Title: The Effect Of The Spiritual Diary On Anxiety and Spiriutal Well-Being In Children Diagnosed With Type1 Diabetes
Brief Title: The Effect Of The Spiritual Diary In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tugce atak meric, Nurse, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: B-TUGCEATAKMERİC-001
Record Dates: First submitted 2022-01-21; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: spirituality; children; anxiety
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There will be three groups in the study. Spiritual Diary Group will be asked to keep a spiritual diary "What Did You Feel Today? The children in Diary Gruop will be asked to keep a diary of "What did You do today? 3 days a week for 4 weeks, and Control Group will be the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spiritual Diary Group (Experimental): -What did you feel today? Spiritual Diary: According to the randomization, the participants in Cluster 1 were asked to write their bad/good memories about the four elements (self, others/family, nature, God/God) in John Fisher's Four Domains model, ask family, others, and God/ God was asked to write down his wishes and wishes, and the child in this group generally wrote the question "What did I feel today?" in his diary.
  Interventions: Other: Diary
- Diary Group (Experimental): What Did You Do Today? Diary: According to randomization, the children in the Cluster 2 group were asked to write down their daily activities and activities (eating, watching TV, time spent with their friends at school, etc.) and the children in this group were asked to generally ask, "What did I do today?" answered the question.
  Interventions: Other: Diary
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Other: Diary — spiritual diary group and diary gruop will write a diary
  Other Names: writing a diary
  Arms: Diary Group; Spiritual Diary Group

SUMMARY:
The research will be carried out in two phases in order to verify the Turkish validity and reliability of the "Feeling Good, Living Life" (FGLL) Scale and to determine the effect of the diary kept using the spiritual writing technique on the anxiety and spiritual well-being level of the children aged 9-12 years who have been diagnosed with Type 1 Diabetes. The first phase of the research was carried out methodologically in Kartal Yavuz Selim Secondary School and Kartal Borsa Imam Hatip Secondary School in Kartal District of Istanbul Province between November-December 2021 for the Turkish validity and reliability study of the FGLL Scale. It has been determined that FGLL can be used as a valid and reliable tool for children aged 9-12 in Turkish society. In the second phase of the study, it was decided to conduct it at Kartal Dr. Lütfi Kırdar City Hospital in order to reach children between the ages of 9 and 12 who were diagnosed with Type 1 Diabetes, and necessary permissions were obtained from the institutions. Istanbul/Kartal Dr. Sample calculations were made with the G*Power 3.1 program in children diagnosed with Type 1 Diabetes, who applied to the Lütfi Kırdar City Hospital Pediatric Endocrinology and Metabolic Diseases Outpatient Clinic. It was calculated that a total of 89 people in three groups, 28/30 people in the groups, should be reached (n=89). The data in the second phase of the study were "Introductory Information Form for Children Diagnosed with Type 1 Diabetes", "Feeling Good-Living Life Scale" and "State-Trait Anxiety Inventory for Children", "What Did You Feel Today? Spiritual Diary" and "What Did You Do Today?Diary" It will be obtained through.

DETAILED DESCRIPTION:
Inclusion Criteria:

Age range of 9-12, Diagnosed with Type 1 Diabetes at least one year ago, Having no other physiological or psychological diseases, No mental disability Does not use psychoactive drugs, Speaking and understanding Turkish, Able to read and write Parents who volunteer their child to participate in the research and sign the consent form, Children in good physical condition were included in the study.

Exclusion Criteria:

Age range not 9-12, Diagnosed with Type 1 Diabetes for less than a year, Having other physiological and psychological diseases, Mentally disabled, Using psychoactive drugs, Can't speak or understand Turkish, illiterate, Parents who do not volunteer for the child to participate in the research, Children who were not in good physical time and had pain were not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 9-12,
* Diagnosed with Type 1 Diabetes at least one year ago,
* Having no other physiological or psychological diseases,
* No mental disability
* Does not use psychoactive drugs,
* Speaking and understanding Turkish,
* Able to read and write
* Parents who volunteer their child to participate in the research and sign the consent form,
* Children in good physical condition were included in the study.

Exclusion Criteria:

* Age range not 9-12,
* Diagnosed with Type 1 Diabetes for less than a year,
* Having other physiological and psychological diseases,
* Mentally disabled,
* Using psychoactive drugs,
* Can't speak or understand Turkish,
* illiterate,
* Parents who do not volunteer for the child to participate in the research,
* Children who were not in good physical time and had pain were not included in the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Spritual well-being | 4 weeks
  Children's spiritual well-being will be evaluated with Feeling Good Living Life Scale
Anxiety | 4 weeks
  Chilren's anxiety level will be evaluated with State-trait Anxiety Invetory for Children

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parilakova M, Babincak P. Feeling Good, Living Life: Evaluation of Psychometric Properties of the Slovak Version in Children Age 8-11 Years. J Relig Health. 2020 Jun;59(3):1421-1433. doi: 10.1007/s10943-019-00867-x. PMID 31250163